CLINICAL TRIAL: NCT01387022
Title: Open Label Randomized Controlled Trial to Assess the Impact of Prophylactic Exposure to Tenofovir Gel on the Efficacy of Subsequent Tenofovir-containing Antiretroviral Therapy on Viral Suppression
Brief Title: Trial to Assess the Impact of PrEP to Tenofovir Gel on the Efficacy of Tenofovir-containing ART on Viral Suppression
Acronym: TOAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for the AIDS Programme of Research in South Africa (Network)
Responsible Party: Principal Investigator, Dr Salim S Abdool Karim, Director, Centre for the AIDS Programme of Research in South Africa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPRISA 009
Record Dates: First submitted 2011-06-21; First posted 2011-07-01 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-03

CONDITIONS: Antiretroviral Treatment Outcomes
Keywords: Antiretroviral treatment; Tenofovir; Drug resistance; Treatment outcome
MeSH Terms: interventions — Tenofovir; Lamivudine; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tenofovir, lamivudine and efavirenz (Experimental)
  Interventions: Drug: Tenofovir, lamivudine and efavirenz
- Zidovudine, lamivudine and efavirenz (Active Comparator)
  Interventions: Drug: Tenofovir, lamivudine and efavirenz

INTERVENTIONS:
Drug: Tenofovir, lamivudine and efavirenz — Tenofovir, 300mg daily, lifelong Lamivudine, 300mg daily, lifelong Efavirenz, 600mg daily, lifelong

SUMMARY:
The HIV/AIDS pandemic remains among the investigators greatest public health challenges. In the absence of an effective vaccine, focus has shifted to other prevention strategies such as pre-exposure prophylaxis. Tenofovir, with potent activity against retroviruses [1], was developed for oral use as Viread®, which is widely used for HIV treatment. The efficacy of Viread® has been demonstrated in treatment-experienced and naïve patients [2,3]. In antiretroviral-naive patients, the combination of tenofovir with lamivudine and efavirenz has been classified as a preferred regimen in the Department of Health and Human Services treatment guidelines[4], and has been adopted by the South African Department of health as the first line regimen in treatment-naïve HIV infected patients since April 2010. The durability of antiviral response, favourable resistance profile, once daily dosing, and excellent long term safety profile of tenofovir [5], makes this drug an attractive option in both treatment and prevention regimens and its long half-life [6], made it an ideal choice as the first antiretroviral drug to be formulated as a microbicide gel.

The CAPRISA 004 study conducted in South Africa which tested the effectiveness and safety of 1% tenofovir gel showed that the use of tenofovir in a gel formulation reduced HIV acquisition by 39% overall, and by 54% in women with high gel adherence [7]. There have been concerns raised regarding the use of tenofovir in both PrEP and treatment regimens due to the potential for selection of viral mutations and development of resistance in patients who have become HIV-infected while on PrEP.

There have been no studies conducted to determine whether using tenofovir in pre-exposure prophylaxis affects treatment outcomes in patients who later use tenofovir, which is part of the first line ART of South Africa.

This study aims to determine whether prophylactic exposure to tenofovir gel alters the therapeutic response to a tenofovir containing antiretroviral regimen.

DETAILED DESCRIPTION:
Purpose:

To determine whether prophylactic exposure to tenofovir gel alters the therapeutic response to a tenofovir containing antiretroviral regimen

Study design:

Open label, two-arm, randomised controlled trial

Study population:

Women who become infected with HIV while participating in the CAPRISA 004 and CAPRISA 008 trials. There are 3 study populations:

Study population 1:

HIV positive women from the CAPRISA 004 tenofovir gel arm and HIV positive women from the clinical trial tenofovir gel provision arm of CAPRISA 008

Study population 2:

HIV positive women in the placebo arm of CAPRISA 004

Study population 3:

HIV positive women from the family planning service arm of CAPRISA 008

Study sites:

CAPRISA eThekwini and CAPRISA Vulindlela clinics.

Study duration:

3 years

Study intervention:

Enrolled women will be initiated on their assigned antiretroviral therapy regimen when they reach any of the following criteria:

* reach a CD4+ count of less than 350 cell/mm3
* acquire an AIDS defining illness
* become pregnant - women in any of the three study populations who become pregnant during follow-up will be initiated on their assigned treatment regimen, as appropriate, for prevention of mother-to-child transmission of HIV.

At enrolment women in each of the three study populations will be assigned randomly to one of the two following antiretroviral regimens Intervention Arm: Tenofovir, lamivudine and efavirenz Control arm: Zidovudine, lamivudine and efavirenz

Sample size: The projected sample size is 90 women. The number of women in each stratum is as follows:

Study population 1: n = 40 Study population 2: n = 30 Study population 3: n = 20

Primary endpoint:

The primary endpoint is the antiretroviral treatment failure rate at 12 months. Treatment failure is defined as viral load > 50 copies/ml, antiretroviral regimen changes for treatment failure or death

Secondary Endpoints:

1. Change in CD4+ cell count from the earliest post-infection timepoint to the time of randomisation to 12, 24 and 36 months post-randomisation
2. Tenofovir resistance, defined as presence of K65R, K70E or any of the TAMS mutations.
3. Reported adverse events with severity grades 3 and 4 based on the DAIDS toxicity grading tables
4. Cellular and humoral immune responses
5. Genital viral shedding (viral load on tear flow) Ancillary Endpoint Mother-to-child HIV transmission rates as determined by PCR on infant at 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Previously enrolled in the CAPRISA 004 or CAPRISA 008 study - placebo or active arms
* Able and willing to provide informed consent to be screened for, and to enrol in, the study
* Able and willing to provide adequate locator information for study retention purposes
* Confirmed HIV infection in the CAPRISA 004 or 008 trial
* Agree to adhere to study visits and procedures

Exclusion Criteria:

* Currently on antiretroviral therapy (including PMTCT prophylaxis)
* Has any other condition that, based on the opinion of the Investigator or designee, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nivashnee Naicker, MBChB, Principal Investigator — Centre for the AIDS Programme of Research in South Africa
Locations (1):
- CAPRISA, Durban, KwaZulu-Natal, South Africa

REFERENCES:
- [Background] De Clercq E. Acyclic nucleoside phosphonates: past, present and future. Bridging chemistry to HIV, HBV, HCV, HPV, adeno-, herpes-, and poxvirus infections: the phosphonate bridge. Biochem Pharmacol. 2007 Apr 1;73(7):911-22. doi: 10.1016/j.bcp.2006.09.014. Epub 2006 Sep 19. PMID 17045247
- [Background] Schooley RT, Ruane P, Myers RA, Beall G, Lampiris H, Berger D, Chen SS, Miller MD, Isaacson E, Cheng AK; Study 902 Team. Tenofovir DF in antiretroviral-experienced patients: results from a 48-week, randomized, double-blind study. AIDS. 2002 Jun 14;16(9):1257-63. doi: 10.1097/00002030-200206140-00008. PMID 12045491
- [Background] Squires K, Pozniak AL, Pierone G Jr, Steinhart CR, Berger D, Bellos NC, Becker SL, Wulfsohn M, Miller MD, Toole JJ, Coakley DF, Cheng A; Study 907 Team. Tenofovir disoproxil fumarate in nucleoside-resistant HIV-1 infection: a randomized trial. Ann Intern Med. 2003 Sep 2;139(5 Pt 1):313-20. doi: 10.7326/0003-4819-139-5_part_1-200309020-00006. PMID 12965939
- [Background] Panel on Antiretroviral Guidelines for Adults and Adolescents. Guidelines for the use of antiretroviral agents in HIV-1-infected adults and adolescents. Guidelines for the use of antiretroviral agents in HIV-1-infected adults and adolescents. December 1, 2009. Available from: www.aidsinfo.nih.gov/contentfiles/AdultandAdolescentGL.pdf. Accessed 9 November 2010.
- [Background] Gallant JE, Staszewski S, Pozniak AL, DeJesus E, Suleiman JM, Miller MD, Coakley DF, Lu B, Toole JJ, Cheng AK; 903 Study Group. Efficacy and safety of tenofovir DF vs stavudine in combination therapy in antiretroviral-naive patients: a 3-year randomized trial. JAMA. 2004 Jul 14;292(2):191-201. doi: 10.1001/jama.292.2.191. PMID 15249568
- [Background] Rohan LC, Moncla BJ, Kunjara Na Ayudhya RP, Cost M, Huang Y, Gai F, Billitto N, Lynam JD, Pryke K, Graebing P, Hopkins N, Rooney JF, Friend D, Dezzutti CS. In vitro and ex vivo testing of tenofovir shows it is effective as an HIV-1 microbicide. PLoS One. 2010 Feb 19;5(2):e9310. doi: 10.1371/journal.pone.0009310. PMID 20174579
- [Background] Abdool Karim Q, Abdool Karim SS, Frohlich JA, Grobler AC, Baxter C, Mansoor LE, Kharsany AB, Sibeko S, Mlisana KP, Omar Z, Gengiah TN, Maarschalk S, Arulappan N, Mlotshwa M, Morris L, Taylor D; CAPRISA 004 Trial Group. Effectiveness and safety of tenofovir gel, an antiretroviral microbicide, for the prevention of HIV infection in women. Science. 2010 Sep 3;329(5996):1168-74. doi: 10.1126/science.1193748. Epub 2010 Jul 19. PMID 20643915
- [Derived] Naicker N, Naidoo A, Werner L, Garrett N, Majola N, Asari V, Baxter C, Grobler A, Karim QA, Karim SSA. Efficacy and safety of tenofovir-containing antiretroviral therapy in women who acquired HIV while enrolled in tenofovir gel prophylaxis trials. Antivir Ther. 2017;22(4):287-293. doi: 10.3851/IMP3106. Epub 2016 Nov 4. PMID 27835613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two arm, open-label, randomised controlled trial
Pre-assignment Details: A total of 214 participants were assessed for eligibility: 60 were excluded due to high CD4+ count, 30 were already on ART, 8 were loss to follow-up and 43 refused participation. Of the 73 that were screened, 8 were screen failures due to high CD4+ count, 4 refused participation, 1 was very ill with TB and 1 could not be contacted.
Groups:
- Tenofovir-containing Regimen: Patients were initiated on EFV, FTC/3TC,TDF
- Tenofovir-sparing Regimen: Patients were initiated on EFV,FTC/3TC,ZDV
Period: Overall Study
Arm/Group | Tenofovir-containing Regimen | Tenofovir-sparing Regimen
Started | 29 | 30
Completed | 28 | 26
Not Completed | 1 | 4
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Population: All participants who were randomised and initiated on ART
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenofovir-containing Regimen | Tenofovir-sparing Regimen | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 28 [25 to 33] | 28 [26 to 30] | 28 [25 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 30 | 59
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 30 | 59
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 29 | 30 | 59
CD4+ T cell count [Median (Inter-Quartile Range); unit: cells/uL] | 345 [289 to 431] | 335 [280 to 411] | 345 [280 to 423]
Viral load [Mean (Standard Deviation); unit: log10 copies/ml] | 4.4 (0.79) | 4.6 (0.80) | 4.5 (0.79)

OUTCOME MEASURES:

1. Primary Outcome: The Antiretroviral Treatment Failure Rate at 12 Months.
Description: Treatment failure is defined as viral load > 50 copies/ml, antiretroviral regimen changes for treatment failure or death
Time Frame: 12 months post ART intiation or until time of death
Population: All participants who randomised and initiated on ART
Measure: Number; unit: participants
Arm/Group | Tenofovir-containing Regimen | Tenofovir-sparing Regimen
Number analyzed (Participants) | 29 | 30
participants | 4 | 5
Statistical Analysis 1: Comparison: Tenofovir-containing Regimen vs Tenofovir-sparing Regimen; Test type: Superiority or Other; p = 1.00, Fisher Exact

2. Secondary Outcome: Change in CD4+ Cell Count From Randomisation to 12 Months Post-randomisation
Description: Difference between 12 months and randomisation CD4+ count was calculated and then summarised
Time Frame: Measured at 12 months post ART initiation
Population: All participants for whom CD4+ count measurements were recorded at randomisation and at 12 months
Measure: Median (Inter-Quartile Range); unit: cells/uL
Arm/Group | Tenofovir-containing Regimen | Tenofovir-sparing Regimen
Number analyzed (Participants) | 21 | 19
cells/uL | 217 [52 to 272] | 174 [70 to 404]
Statistical Analysis 1: Comparison: Tenofovir-containing Regimen vs Tenofovir-sparing Regimen; Test type: Superiority or Other; p = 0.481, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Tenofovir Resistance, Defined as Presence of K65R, K70E or Any of the TAMS Mutations
Time Frame: From randomisation until either time of termination or time of death
Population: Resistance testing was only done on participants who were failing first line antiretroviral therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir-containing Regimen | Tenofovir-sparing Regimen
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

4. Secondary Outcome: Reported Adverse Events With Severity Grades 3 and 4 Based on the DAIDS Toxicity Grading Tables
Time Frame: From randomisation until either time of termination or time of death
Population: All participants who randomised and initiated on ART
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir-containing Regimen | Tenofovir-sparing Regimen
Number analyzed (Participants) | 29 | 30
Participants | 7 | 12
Statistical Analysis 1: Comparison: Tenofovir-containing Regimen vs Tenofovir-sparing Regimen; Test type: Superiority or Other; p = 0.267, Fisher Exact

5. Secondary Outcome: Cellular and Humoral Immune Responses
Description: We will assess whether exposure to tenofovir gel at the time of HIV acquisition alters the subsequent humoral and cellular immune responses following antiretroviral treatment initiation
Time Frame: 3 years
Population: Data were not collected for this Outcome Measure
Arm/Group | Tenofovir-containing Regimen | Tenofovir-sparing Regimen
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Genital Viral Shedding (Viral Load on Tear Flow)
Time Frame: 3 years
Population: Data were not collected for this Outcome Measure
Arm/Group | Tenofovir-containing Regimen | Tenofovir-sparing Regimen
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 19 July 2011 to 30 September 2014
Arm/Group | Tenofovir-containing Regimen | Tenofovir-sparing Regimen
Serious Adverse Events (participants affected / at risk) | 10/29 | 11/30
Other Adverse Events (participants affected / at risk) | 1/29 | 5/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenofovir-containing Regimen (N=29) | Tenofovir-sparing Regimen (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 1 (1) | 0 (0)
Hyperlactacidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Delivery (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 1 (1)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Abscess drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Caesarean section (Surgical and medical procedures) | 2 (2) | 3 (3)
Female sterilisation (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tenofovir-containing Regimen (N=29) | Tenofovir-sparing Regimen (N=30)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bartholin's abscess (Infections and infestations) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The main limitation of the study was the small sample size. The eligible pool of participants was dependent on two other tenofovir gel trials, one of which experienced long delay in starting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No